CLINICAL TRIAL: NCT04888702
Title: Holter of Movement in Patients with Type 2 or 3 Spinal Muscular Atrophy When Initiating Treatment with Spinraza ° or Risdiplam. Acti-SMA Study.
Brief Title: Holter of Movement in Patients with SMA Undergoing Treatment.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Collaborators: SYSNAV (Industry); Erasme University Hospital (Other); Queen Fabiola Children's University Hospital (Other); Centre Hospitalier Régional de la Citadelle (Other)
Responsible Party: Principal Investigator, Margaux POLEUR, Doctor, Centre Hospitalier Universitaire de Liege
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ActiSMA.
Record Dates: First submitted 2021-03-11; First posted 2021-05-17 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-05

CONDITIONS: Spinal Muscular Atrophy
Keywords: Actimyo; Accelerometry; Motor neuron disease; Risdiplam; Nusinersen; Home monitoring
MeSH Terms: conditions — Muscular Atrophy, Spinal; Motor Neuron Disease

STUDY DESIGN:
Intervention Model Description: all patients undergo clinical evaluation and wear Actimyo device in daily living to evaluate their improvement under treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SMA patients (Experimental): Patients with type 2 or 3 spinal muscular atrophy undergoing Spinraza° or risdiplam treatment.
  Interventions: Device: Actimyo

INTERVENTIONS:
Device: Actimyo — Actimyo° is an innovative device intended to be used in a home-based environment. It is composed of two watch-like sensors, each containing a magneto-inertial sensors that record the linear acceleration, the angular velocity, the magnetic field of the movement in all directions.The two watches can be worn as wristwatch or placed near the ankle.

SUMMARY:
Acti-SMA is a multi-centric academic study. It aims to monitor the progress of patients with spinal muscular atrophy under treatment with Spinraza° or risdiplam. First, we want to quantify improvement of both ambulant and non-ambulant patients under treatment. A secondary objective would also be to identify suitable accelerometric measurements that are sensitive to change but also well correlated to other clinical scores.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed spinal muscular atrophy.
* Treatment by Spinraza ° or by risdiplam planned.
* Over 6 years old.
* Signed informed consent.

Exclusion Criteria:

- Patients with excessive cognitive disorders, limiting the understanding of task or with apparent communication difficulties hindering data collection.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-08-08 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
95th centile of stride velocity | 39 months
  95th centile of stride velocity obtained with a magneto-inertial sensor (Actimyo°) in real-life.
  (meter per second).
50th centile of stride velocity | 39 months
  50th centile of stride velocity obtained with a magneto-inertial sensor (Actimyo°) in real-life (meter per second).
95th centile of stride length | 39 months
  95th centile of stride length obtained with a magneto-inertial sensor (Actimyo°) in real-life (meter).
50th centile of stride length | 39 months
  50th centile of stride length obtained with a magneto-inertial sensor (Actimyo°) in real-life (meter).
Upper limb function evolution in patient with SMA undergoing treatment | 39 months
  Upper limb function assessed with a magneto-inertial sensor (Actimyo°) in real-life.

SECONDARY OUTCOMES:
6-minute walk test | 39 months
  The Six-Minute Walk Test is a functional walking test in which investigators assess the distance the patient can walk in six minutes (meter).
Dynamometric measures | 39 months
  Assessment of upper limb strength with myogrip and myopinch (kg).
10-metre walk test | 39 months
  The 10-metre walk test is a functional walking test in which investigators assess the time the patient take to walk 10 meters (second).
rise from floor | 39 months
  The rise from floor is a functional test in which investigators assess the time the patient take to rise from the floor (second).
4-stair climb | 39 months
  The 4-stair climbr is a functional test in which investigators assess the time the patient take to climb a four-step staircase (second).
revised upper limb module (RULM) | 39 months
  Revised Upper Limb Module (RULM) is an assessment specifically designed for upper limb function in Spinal Muscular Atrophy.
Hamersmith funcitonnal motor scale (HFMS) | 39 months
  HFMS is a scale is specifically designed outcome measure for people affected by Spinal Muscular Atrophy.
motor function measure (MFM) | 39 months
  Motor Function Measure is a global quantitative scale created to measure the functional motor abilities of a person affected by a neuromuscular disease.

CONTACTS AND LOCATIONS:
Overall Officials: Margaux Poleur, Principal Investigator — CHR Citadelle-CHU liège
Locations (3):
- Belgium (2):
  - Centre Hospitalier Régional de la Citadelle, Liège, Liège
  - Erasme Hospital - Cliniques universitaires de Bruxelles, Brussels
- National Clinical Hospital for Children Neurohabilitation "Dr Nicolae Robanescu", Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No